CLINICAL TRIAL: NCT00823082
Title: A Prospective Randomized Pilot Study to Evaluate the Effect of Preoperative Antithrombin Supplementation on Postoperative Levels of Antithrombin in Patients Undergoing Cardiac Surgery With Cardiopulmonary Bypass
Brief Title: Use of Antithrombin in Cardiac Surgery With Cardiopulmonary Bypass
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Instituto Grifols, S.A. (Industry)
Responsible Party: Sponsor
Organization: Grifols Biologicals, LLC (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IG0801
Record Dates: First submitted 2009-01-14; First posted 2009-01-15 (Estimated); Results first posted 2016-08-04 (Estimated); Last update posted 2016-09-20 (Estimated); Status verified 2016-08

CONDITIONS: Acquired Antithrombin III Deficiency; Coronary Artery Bypass
Keywords: antithrombin; ATIII; acquired deficiency; anticoagulants; cardiopulmonary bypass; surgery; complications; postoperative outcomes
MeSH Terms: interventions — Antithrombin III

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Antithrombin III treatment group (Experimental): Preoperative ATIII supplementation administered immediately after anesthesia induction
  Interventions: Drug: Antithrombin III
- Control group (No Intervention): No preoperative ATIII supplementation administered

INTERVENTIONS:
Drug: Antithrombin III — Single dose of antithrombin III sufficient to achieve a preoperative level of 120%
  Other Names: Anbinex; ATIII
  Arms: Antithrombin III treatment group

SUMMARY:
The purpose of this trial is to study the effects of preoperative antithrombin supplementation in patients undergoing cardiac surgery with cardiopulmonary bypass in order to maintain antithrombin levels in a range greater than 58% of functional activity and, eventually, to decrease negative clinical outcomes during the ICU stay.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* At least 18 years of age
* Subject needed elective cardiac surgery with cardiopulmonary bypass except for heart transplantation
* Subject had a baseline ATIII level of less than 100% and equal to or above 60%
* Subject signed the informed consent form
* Subject was willing to comply with all aspects of the protocol, including blood sampling, for the total duration of the study

Exclusion Criteria:

* Documented congenital ATIII deficiency or ATIII levels below 60%
* Subject had a baseline ATIII level of 100% or higher
* Subject needed emergency (non-elective) surgery
* Subject needed heart transplantation
* History of anaphylactic reaction(s) to blood or blood components
* Allergies to excipients
* Subject was pregnant
* Subject had any medical condition that according to the investigators judgment worsens the surgical outcome above the expected
* Subject had any medical condition which is likely to interfere with the evaluation of the study treatment and/or the satisfactory conduct of the trial according to the investigators judgment
* Subject had participated in any another investigational study within the last 30 days previous to the inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2009-06; Primary Completion 2011-06 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marco Ranucci, MD, Principal Investigator — IRCCS Policlinico San Donato, Milano
Locations (1):
- IRCCS Policlinico San Donato, Milan, Lombardy, Italy

REFERENCES:
- [Derived] Ranucci M, Baryshnikova E, Crapelli GB, Woodward MK, Paez A, Pelissero G. Preoperative antithrombin supplementation in cardiac surgery: a randomized controlled trial. J Thorac Cardiovasc Surg. 2013 May;145(5):1393-9. doi: 10.1016/j.jtcvs.2012.09.061. Epub 2012 Oct 25. PMID 23102903

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Antithrombin III Treatment Group | Control Group
Started | 100 | 100
Safety Population | 100 | 99
Intent-to-Treat/Per Protocol Populations | 100 | 94
Completed | 100 | 99
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Population: 206 subjects were randomized; six were screen failures. 100 subjects in the Anbinex treatment group and 94 subjects in the control group were included in the Intent-to-treat and Per-protocol populations (6 subjects in the control group were excluded). 199 subject were included in the Safety population (100 Anbinex and 99 control).
Groups:
- Total: Total of all reporting groups
Arm/Group | Antithrombin III Treatment Group | Control Group | Total
Number analyzed (Participants) | 100 | 94 | 194
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.51 (10.48) | 67.63 (11.18) | 67.05 (10.81)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 24 | 41
  Male | 83 | 70 | 153
Region of Enrollment [Number; unit: participants]
  Italy | 100 | 94 | 194

OUTCOME MEASURES:

1. Primary Outcome: Postoperative ATIII Levels at the ICU Admission
Description: Measurement of postoperative ATIII functional activity at ICU admission
Time Frame: ICU admission
Population: Intent-to-treat set and Per-protocol set
Measure: Mean (Standard Deviation); unit: IU
Arm/Group | Antithrombin III Treatment Group | Control Group
Number analyzed (Participants) | 100 | 94
IU | 94.06 (13.74) | 64.70 (9.89)
Statistical Analysis 1: Comparison: Antithrombin III Treatment Group vs Control Group; Test type: Superiority or Other; p < 0.0001, ANCOVA

2. Primary Outcome: Percentage of Subjects With ATIII Levels of 58% or Higher at ICU Admission
Description: Percentage of subjects with ATIII levels of 58% functional activity or higher at ICU admission
Time Frame: ICU admission
Population: Intent-to treat set and Per-protocol set
Measure: Number; unit: percentage of participants
Arm/Group | Antithrombin III Treatment Group | Control Group
Number analyzed (Participants) | 100 | 94
percentage of participants | 100.0 | 74.5
Statistical Analysis 1: Comparison: Antithrombin III Treatment Group vs Control Group; Test type: Superiority or Other; p < 0.0001, Fisher Exact

3. Secondary Outcome: Percentage of Subjects With Postoperative Myocardial Infarction
Description: Percentage of subjects with postoperative myocardial infarction defined through enzymatic criteria plus new Q-waves at the electrocardiogram
Time Frame: During ICU stay (maximum 70 days)
Population: Intent-to-treat set
Measure: Number; unit: percentage of participants
Arm/Group | Antithrombin III Treatment Group | Control Group
Number analyzed (Participants) | 100 | 94
percentage of participants
  Follow-up visit (Anbinex n=76, Control n=69) | 0.0 | 0.0
  ICU discharge visit (Anbinex n=99, Control n=93) | 1.0 | 2.2
Statistical Analysis 1: Comparison: Antithrombin III Treatment Group vs Control Group; At ICU discharge visit; Test type: Superiority or Other; p = 0.6115, Fisher Exact

4. Secondary Outcome: Percentage of Subjects With Adverse Neurologic Outcome
Description: Percentage of subjects with adverse neurologic outcome defined as: coma, stroke or psychotic behaviors lasting >12 hours after extubation
Time Frame: During ICU stay (maximum 70 days)
Population: Intent-to-treat set
Measure: Number; unit: percentage of participants
Arm/Group | Antithrombin III Treatment Group | Control Group
Number analyzed (Participants) | 100 | 94
percentage of participants
  Follow-up visit (Anbinex n=75, Control n=69) | 5.3 | 0.0
  ICU discharge visit (Anbinex n=99, Control n=93) | 1.0 | 0.0
Statistical Analysis 1: Comparison: Antithrombin III Treatment Group vs Control Group; Follow-up visit; Test type: Superiority or Other; p = 0.1211, Fisher Exact
Statistical Analysis 2: Comparison: Antithrombin III Treatment Group vs Control Group; ICU discharge visit; Test type: Superiority or Other; p = 1.000, Fisher Exact

5. Secondary Outcome: Percentage of Patients With Thromboembolic Events
Description: Percentage of subjects with thromboembolic events defined as perioperative myocardial infarction, stroke, mesenteric infarction, peripheral thromboembolism and pulmonary embolism
Time Frame: During ICU stay (maximum 70 days)
Population: Intent-to-treat set
Measure: Number; unit: percentage of participants
Arm/Group | Antithrombin III Treatment Group | Control Group
Number analyzed (Participants) | 100 | 94
percentage of participants
  Follow-up visit (Anbinex n=76, Control n=69) | 0.0 | 0.0
  ICU discharge visit (Anbinex n=99, Control n=94) | 0.0 | 1.1
Statistical Analysis 1: Comparison: Antithrombin III Treatment Group vs Control Group; ICU discharge visit; Test type: Superiority or Other; p = 0.4870, Fisher Exact

6. Secondary Outcome: ICU Stay Duration
Time Frame: During ICU stay (maximum 70 days)
Population: Intent-to-treat set. One subject in the control group was missing this data.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Antithrombin III Treatment Group | Control Group
Number analyzed (Participants) | 100 | 93
days | 2.00 [1.00 to 4.00] | 2.00 [1.00 to 3.00]
Statistical Analysis 1: Comparison: Antithrombin III Treatment Group vs Control Group; Test type: Superiority or Other; p = 0.3897, Hodges-Lehmann test

7. Secondary Outcome: In-hospital Postoperative Mortality
Time Frame: 70 days after ICU admission (maximum)
Population: Intent-to-treat set. One subject in the control group was missing this data.
Measure: Number; unit: percentage of participants
Arm/Group | Antithrombin III Treatment Group | Control Group
Number analyzed (Participants) | 100 | 93
percentage of participants | 1.0 | 1.1
Statistical Analysis 1: Comparison: Antithrombin III Treatment Group vs Control Group; Test type: Superiority or Other; p = 1.0000, Fisher Exact

8. Secondary Outcome: Heparin Resistance
Description: Percentage of subjects with heparin resistance defined as failure to reach an activated clotting time >450 seconds after a dose of up to 400 IU/kg of heparin, or failure to maintain this activated clotting time value despite heparin supplementations of 100 IU/kg per each dose with an interval of at least 30 minutes between doses
Time Frame: Immediately after anesthesia induction
Population: Intent-to-treat set. One subject in the Antithrombin III treatment group was missing this data.
Measure: Number; unit: percentage of participants
Arm/Group | Antithrombin III Treatment Group | Control Group
Number analyzed (Participants) | 99 | 94
percentage of participants | 17.2 | 40.4
Statistical Analysis 1: Comparison: Antithrombin III Treatment Group vs Control Group; Test type: Superiority or Other; p = 0.0004, Fisher Exact

9. Secondary Outcome: Postoperative Blood Loss in First 12 Hours
Description: Blood loss defined as the amount of blood collected in the cardiotomy reservoir from ICU admission through the following 12 hours
Time Frame: ICU admission through 12 hours post-operative
Population: Intent-to-treat set. One subject in the Antithrombin III treatment group was missing this data.
Measure: Least Squares Mean (Standard Error); unit: mL
Arm/Group | Antithrombin III Treatment Group | Control Group
Number analyzed (Participants) | 99 | 94
mL | 516.11 (30.292) | 415.00 (31.087)
Statistical Analysis 1: Comparison: Antithrombin III Treatment Group vs Control Group; Test type: Superiority or Other; p = 0.0209, ANCOVA

10. Secondary Outcome: Need for Blood Products
Description: Number of units of packed red blood cells, fresh frozen plasma, and/or platelets needed
Time Frame: During ICU stay (maximum 70 days)
Population: Intent-to-treat set
Measure: Least Squares Mean (Standard Error); unit: Units
Arm/Group | Antithrombin III Treatment Group | Control Group
Number analyzed (Participants) | 100 | 94
Units
  Packed Red Blood Cells (Anbinex n=45,Control n=38) | 43.711 (3.551) | 41.987 (3.864)
  Fresh frozen plasma (Anbinex n=16, Control n=8) | 12.188 (1.646) | 13.125 (2.327)
  Platelets (Anbinex n=5, Control n=8) | 8.500 (1.564) | 6.188 (1.236)
Statistical Analysis 1: Comparison: Antithrombin III Treatment Group vs Control Group; Number of units of packed red blood cells; Test type: Superiority or Other; p = 0.7433, ANCOVA
Statistical Analysis 2: Comparison: Antithrombin III Treatment Group vs Control Group; Units of fresh frozen plasma; Test type: Superiority or Other; p = 0.7453, ANCOVA
Statistical Analysis 3: Comparison: Antithrombin III Treatment Group vs Control Group; Units of platelets; Test type: Superiority or Other; p = 0.2705, ANCOVA

11. Secondary Outcome: Percentage of Subjects Needing Surgical Re-exploration
Description: Percentage of subjects needing surgical re-exploration resulting from bleeding
Time Frame: During ICU stay (maximum 70 days)
Population: Intent-to-treat set. Two subjects in the Antithrombin III treatment group and 2 subjects in the Control group were missing this data.
Measure: Number; unit: percentage of participants
Arm/Group | Antithrombin III Treatment Group | Control Group
Number analyzed (Participants) | 98 | 92
percentage of participants | 5.1 | 2.2
Statistical Analysis 1: Comparison: Antithrombin III Treatment Group vs Control Group; Test type: Superiority or Other; p = 0.4460, Fisher Exact

12. Secondary Outcome: Percentage of Subjects With Low Cardiac Syndrome
Description: Percentage of subjects with low cardiac syndrome defined as the need for major inotropic support or intra-aortic balloon pump
Time Frame: During ICU stay (maximum 70 days)
Population: Intent-to-treat set. Three subjects in the Antithrombin III treatment group and 1 subject in the Control group were missing this data.
Measure: Number; unit: percentage of participants
Arm/Group | Antithrombin III Treatment Group | Control Group
Number analyzed (Participants) | 97 | 93
percentage of participants | 24.7 | 20.4
Statistical Analysis 1: Comparison: Antithrombin III Treatment Group vs Control Group; Test type: Superiority or Other; p = 0.4936, Fisher Exact

13. Secondary Outcome: Percentage of Subjects With Renal Dysfunction
Description: Percentage of subjects with renal dysfunction defined as an increase of serum creatinine levels to >2.0 and twice the baseline level or need for renal replacement therapy
Time Frame: During ICU stay (maximum 70 days)
Population: Intent-to-treat set
Measure: Number; unit: Percentage of participants
Arm/Group | Antithrombin III Treatment Group | Control Group
Number analyzed (Participants) | 100 | 94
Percentage of participants
  Follow-up visit (Anbinex n=75, Control n=69) | 1.3 | 0.0
  ICU discharge visit (Anbinex n=99, Control n=93) | 3.0 | 1.1
Statistical Analysis 1: Comparison: Antithrombin III Treatment Group vs Control Group; Follow-up visit; Test type: Superiority or Other; p = 1.000, Fisher Exact
Statistical Analysis 2: Comparison: Antithrombin III Treatment Group vs Control Group; ICU discharge visit; Test type: Superiority or Other; p = 0.6218, Fisher Exact

14. Secondary Outcome: Mechanical Ventilation Duration
Time Frame: During ICU stay (maximum 70 days)
Population: Intent-to-treat set
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Antithrombin III Treatment Group | Control Group
Number analyzed (Participants) | 100 | 94
Days | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
Statistical Analysis 1: Comparison: Antithrombin III Treatment Group vs Control Group; Test type: Superiority or Other; p = 0.9574, Hodges-Lehmann

15. Secondary Outcome: Length of Hospital Stay
Description: Length of hospital stay (days) in both groups was defined as the discharge date minus the surgery date plus 1 day, during a maximum of 70 days after ICU admission.
Time Frame: During ICU stay (maximum 70 days)
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Antithrombin III Treatment Group | Control Group
Number analyzed (Participants) | 100 | 94
days | 10.00 [8.00 to 13.50] | 10.00 [8.00 to 13.00]
Statistical Analysis 1: Comparison: Antithrombin III Treatment Group vs Control Group; Test type: Superiority or Other; p = 0.7489, Hodges-Lehmann test

ADVERSE EVENTS:
Time Frame: From the time of the Recruitment Visit (Day -14) to the Follow-up Visit (Day 50 +/- 20 days)
Description: 206 subjects were randomized; six were screen failures. 199 subject were included in the Safety population (100 Anbinex and 99 control).One subject in the control group was excluded from the safety population as Anbinex was administered during the ICU stay.
Groups:
- Control Group: No preoperative ATII supplementation administered
Arm/Group | Antithrombin III Treatment Group | Control Group
Serious Adverse Events (participants affected / at risk) | 32/100 | 29/99
Other Adverse Events (participants affected / at risk) | 96/100 | 97/99
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Antithrombin III Treatment Group (N=100) | Control Group (N=99)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 22 (22) | 17 (17)
Atrial flutter (Cardiac disorders) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 0 (0) | 2 (2)
Cardiac arrest (Cardiac disorders) | 2 (3) | 0 (0)
Cardiac tamponade (Cardiac disorders) | 1 (1) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 2 (2)
Low cardiac output syndrome (Cardiac disorders) | 1 (1) | 3 (3)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular fibrillation (Cardiac disorders) | 0 (0) | 2 (2)
Ventricular hypokinesia (Cardiac disorders) | 0 (0) | 1 (1)
Device occlusion (General disorders) | 0 (0) | 1 (1)
Hyperpyrexia (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Acinetobacter infection (Infections and infestations) | 1 (1) | 0 (0)
Endocarditis (Infections and infestations) | 0 (0) | 1 (1)
Klebsiella infection (Infections and infestations) | 2 (2) | 0 (0)
Pseudomonas infection (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Serratia infection (Infections and infestations) | 1 (1) | 0 (0)
Staphyloccal infection (Infections and infestations) | 1 (1) | 0 (0)
Wound infection Staphyloccal (Infections and infestations) | 0 (0) | 1 (1)
Graft thrombosis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post procedural hemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vasoplegia syndrome (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Wound secretion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Electrocardiogram ST segment elevation (Investigations) | 0 (0) | 1 (1)
Enterococcus test positive (Investigations) | 1 (1) | 0 (0)
Seroconversion test (Investigations) | 1 (1) | 0 (0)
Staphylcoccus test positive (Investigations) | 1 (1) | 0 (0)
Muscle necrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Cerebral hematoma (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral hemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Coma (Nervous system disorders) | 2 (2) | 0 (0)
Psychotic behavior (Psychiatric disorders) | 1 (1) | 0 (0)
Oliguria (Renal and urinary disorders) | 2 (2) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0)
Acute pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Acute respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Evidence based treatment (Surgical and medical procedures) | 0 (0) | 2 (2)
Hospitalization (Surgical and medical procedures) | 0 (0) | 1 (1)
Tricuspid valve repair (Surgical and medical procedures) | 0 (0) | 1 (1)
Hemodynamic instability (Vascular disorders) | 1 (1) | 0 (0)
Hemorrhage (Vascular disorders) | 2 (2) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 1 (1)
Septic shock (Infections and infestations) | 2 (2) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Antithrombin III Treatment Group (N=100) | Control Group (N=99)
Leukocytosis (Blood and lymphatic system disorders) | 12 (12) | 11 (11)
Atrial fibrillation (Cardiac disorders) | 24 (24) | 17 (17)
Atrioventricular block (Cardiac disorders) | 5 (5) | 2 (2)
Bradycardia (Cardiac disorders) | 23 (23) | 12 (12)
Pericardial effusion (Cardiac disorders) | 5 (5) | 5 (5)
Sinus tachycardia (Cardiac disorders) | 4 (4) | 5 (5)
Supraventricular extrasystoles (Cardiac disorders) | 8 (8) | 6 (6)
Tachycardia (Cardiac disorders) | 21 (21) | 17 (17)
Oedema peripheral (General disorders) | 16 (16) | 15 (15)
Pyrexia (General disorders) | 38 (38) | 42 (45)
Serositis (General disorders) | 6 (6) | 5 (5)
Electrocardiogram ST segment elevation (Investigations) | 5 (5) | 4 (4)
Hematocrit decreased (Investigations) | 22 (22) | 6 (7)
Disorientation (Psychiatric disorders) | 6 (6) | 1 (1)
Oliguria (Renal and urinary disorders) | 7 (7) | 2 (2)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 6 (6)
Dyspnoa (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 3 (3)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 10 (10) | 10 (10)
Increased bronchial secretion (Respiratory, thoracic and mediastinal disorders) | 9 (9) | 5 (5)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 47 (47) | 45 (45)
Subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 5 (5) | 0 (0)
Diuretic therapy (Surgical and medical procedures) | 15 (15) | 15 (15)
Hemorrhage (Vascular disorders) | 27 (27) | 23 (23)
Hypertension (Vascular disorders) | 8 (8) | 10 (11)
Hypotension (Vascular disorders) | 11 (11) | 13 (13)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 7 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Site may publish results from the Study, after providing Sponsor thirty days' notice prior to submitting a manuscript or other materials related to the Study to any outside party. At Sponsor's request, Site will remove any Confidential Information (other than Study results), and Site will upon Sponsor's request, delay publication or presentation for a period of up to one hundred twenty days to allow Sponsor to protect its interests in any Sponsor's Inventions.